CLINICAL TRIAL: NCT00709891
Title: Evaluation of the Cobas® 4800 HPV Test for the Detection of High-grade Cervical Disease in Women Undergoing Routine Cervical Cancer Screening
Brief Title: Evaluation of the Cobas® 4800 HPV Test for the Detection of High-grade Cervical Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RD000649; MWP-HPV-159 (Other: Roche Molecular Systems, Inc.)
Record Dates: First submitted 2008-06-30; First posted 2008-07-03 (Estimated); Results first posted 2015-02-09 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Human Papilloma Virus (HPV)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- cobas® 4800 HPV Test (Experimental): The cobas 4800 human papillomavirus (HPV) Test combines in a single assay the identification of pooled high-risk oncogenic HPV types (31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, 68), as well as genotypes 16 and 18 individually.
  Interventions: Device: cobas® 4800 HPV Test

INTERVENTIONS:
Device: cobas® 4800 HPV Test

SUMMARY:
This study provided data on the performance of the Cobas® 4800 HPV Test for identifying histologically confirmed high-grade cervical disease. The baseline, cross-sectional phase was conducted in approximately 45,000 women undergoing routine cervical cancer screening, of whom approximately 7,400 were selected to undergo colposcopy and biopsy/endocervical curettage (ECC) at baseline. These subjects included women with cytology that is 'not normal' and a selection of those with 'normal' cytology who entered a follow-up phase and underwent cytological evaluation annually for 3 years. In this follow-up phase, colposcopy and biopsy/ECC were performed only in women with cervical cytology considered 'not normal' at any of the annual follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 21 years of age presenting for routine cervical cancer screening.
* An intact cervix.
* Willing and able to undergo colposcopy and biopsy and endocervical curettage within 8 weeks after study Visit 1.

Exclusion Criteria:

* Known pregnancy at study Visit 1.
* Presenting for colposcopy at study Visit 1.
* Any condition resulting in increased risk of bleeding at biopsy.
* Hysterectomy.
* Known history of ablative or excisional therapy to the cervix within the preceding 12 months.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47208 (Actual)
Dates: Start 2008-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Behrens, Study Director — Roche Molecular Systems, Inc
Locations (57):
- United States (57):
  - Enterprise, Alabama
  - Hoover, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Carmichael, California
  - Costa Mesa, California
  - Fountain Valley, California
  - San Diego, California
  - Colorado Springs, Colorado
  - Lakewood, Colorado
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Jupiter, Florida
  - Lake Worth, Florida
  - Miami, Florida
  - North Miami, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Decatur, Georgia
  - Roswell, Georgia
  - Boise, Idaho
  - Champaign, Illinois
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Louisville, Kentucky
  - Paducah, Kentucky
  - Covington, Louisiana
  - Ruston, Louisiana
  - Saginaw, Michigan
  - Las Vegas, Nevada
  - Lawrenceville, New Jersey
  - Moorestown, New Jersey
  - Albuquerque, New Mexico
  - New Bern, North Carolina
  - Winston-Salem, North Carolina
  - Englewood, Ohio
  - Lansdale, Pennsylvania
  - West Reading, Pennsylvania
  - Columbia, South Carolina
  - Hilton Head, South Carolina
  - North Charleston, South Carolina
  - Chattanooga, Tennessee
  - Johnson City, Tennessee
  - Nashville, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - McAllen, Texas
  - Temple, Texas
  - Salt Lake City, Utah
  - Virginia Beach, Virginia
  - Tacoma, Washington

REFERENCES:
- [Derived] Monsonego J, Cox JT, Behrens C, Sandri M, Franco EL, Yap PS, Huh W. Prevalence of high-risk human papilloma virus genotypes and associated risk of cervical precancerous lesions in a large U.S. screening population: data from the ATHENA trial. Gynecol Oncol. 2015 Apr;137(1):47-54. doi: 10.1016/j.ygyno.2015.01.551. Epub 2015 Feb 8. PMID 25667973
- [Derived] Wright TC Jr, Stoler MH, Behrens CM, Sharma A, Sharma K, Apple R. Interlaboratory variation in the performance of liquid-based cytology: insights from the ATHENA trial. Int J Cancer. 2014 Apr 15;134(8):1835-43. doi: 10.1002/ijc.28514. Epub 2013 Oct 29. PMID 24122508
- [Derived] Castle PE, Stoler MH, Wright TC Jr, Sharma A, Wright TL, Behrens CM. Performance of carcinogenic human papillomavirus (HPV) testing and HPV16 or HPV18 genotyping for cervical cancer screening of women aged 25 years and older: a subanalysis of the ATHENA study. Lancet Oncol. 2011 Sep;12(9):880-90. doi: 10.1016/S1470-2045(11)70188-7. Epub 2011 Aug 22. PMID 21865084

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had not met the study primary clinical endpoint of ≥ CIN2 were invited to participate in the longitudinal follow-up phase.
Period: Baseline, Cross-sectional Phase
Arm/Group | Cobas® 4800 HPV Test
Started | 47208
Completed | 45758
Not Completed | 1450
Period: Longitudinal Follow-up Phase
Arm/Group | Cobas® 4800 HPV Test
Started | 10002 (Only participants who met study criteria in the Baseline phase started the Follow-up phase.)
Completed | 5020
Not Completed | 4982

BASELINE CHARACTERISTICS:
Population: Eligible population: All participants who met the study inclusion/exclusion criteria, had not been enrolled in the study previously, and had not withdrawn consent before undergoing any study procedures. Of the enrolled population, 321 participants did not meet these criteria.
Arm/Group | Cobas® 4800 HPV Test
Number analyzed (Participants) | 46887
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46887
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Diagnosis of ≥ CIN2
Description: A diagnosis of ≥ CIN2 (cervical intraepithelial neoplasia) included histology results of CIN2, CIN3, adenocarcinoma in situ, squamous cell carcinoma, or adenocarcinoma. The diagnosis was based on central pathology review.
Time Frame: Baseline to the end of the Baseline period (up to 12 weeks)
Population: Evaluable ASC-US participant population: All enrolled participants with a diagnosis of atypical squamous cells of undetermined significance (ASC-US).
Measure: Number; unit: Percentage of participants
Arm/Group | Cobas® 4800 HPV Test
Number analyzed (Participants) | 1578
Percentage of participants
  Positive cobas 4800 HPV test result - n=514 | 14.0
  Negative cobas 4800 HPV test result - n=1064 | 0.8

2. Secondary Outcome: Percentage of Participants With a Diagnosis of ≥ CIN3
Description: A diagnosis of ≥ CIN3 (cervical intraepithelial neoplasia) included histology results of CIN3, adenocarcinoma in situ, squamous cell carcinoma, or adenocarcinoma. The diagnosis was based on central pathology review.
Time Frame: Baseline to the end of the study (up to 5 years, 1 month)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cobas® 4800 HPV Test
Number analyzed (Participants) | 1578
Percentage of participants
  Positive cobas 4800 HPV test result - n=514 | 8.4
  Negative cobas 4800 HPV test result - n=1064 | 0.3

ADVERSE EVENTS:
Description: Safety population: All enrolled participants. Non-serious adverse events were not recorded in this study.
Arm/Group | Cobas® 4800 HPV Test
Serious Adverse Events (participants affected / at risk) | 1/47208
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cobas® 4800 HPV Test (N=47208)
Urogenital haemorrhage (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.